CLINICAL TRIAL: NCT02936752
Title: A Phase 1b Study of the Anti-PD1 Antibody Pembrolizumab in Combination With the Histone Deacetylase Inhibitor, Entinostat for Treatment of Patients With Myelodysplastic Syndromes After DNA Methyltransferase Inhibitor Therapy Failure
Brief Title: Testing the Safety and Efficacy of the Combination of the Antibody Pembrolizumab and Entinostat in Patients With Myelodysplastic Syndrome Who Are Not Responding to Hypomethylating Agents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01501; NCI-2016-01501 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HIC 2000020860; 10009 (Other: Yale University Cancer Center LAO); 10009 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Results first posted 2024-10-01 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — entinostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (entinostat, pembrolizumab) (Experimental): Patients receive lower dose entinostat PO on days 1 and 8 or higher dose entinostat PO on days 1, 8, and 15, and pembrolizumab IV over 30 minutes on day 1 of cycle 2 and cycles thereafter. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve an objective response or maintain a SD status after the first 4 cycles may continue to receive entinostat and pembrolizumab for up to 1 year.
  Interventions: Drug: Entinostat; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS 275; MS-275; MS275; SNDX 275; SNDX-275; SNDX275
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; QL2107; RPH 075; RPH-075; RPH075; SCH 900475; SCH-900475; SCH900475

SUMMARY:
This phase Ib trial studies the side effects and best dose of entinostat when given together with pembrolizumab in treating patients with myelodysplastic syndrome after deoxyribonucleic acid (DNA) methyltransferase inhibitor (DNMTi) therapy failure. Entinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving entinostat together with pembrolizumab may work better in treating patients with myelodysplastic syndrome after DNMTi therapy failure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess safety, tolerability, and identify the maximum tolerated dose (MTD) of entinostat given in combination with MK-3475 (pembrolizumab).

SECONDARY OBJECTIVE:

I. To obtain a preliminary estimate of efficacy of entinostat in combination with MK-3475 (pembrolizumab).

EXPLORATORY OBJECTIVE:

I. To assess the dynamic quantitative change in measurable immunological biomarkers (proportions of myeloid-derived suppressor cells [MDSCs], and programmed death protein-1 [PD-1] expression in bone marrow) with the combined epigenetic-immunotherapy and correlation with any observed clinical responses.

OUTLINE: This is a dose-escalation study of entinostat.

Patients receive lower dose entinostat orally (PO) on days 1 and 8 or higher dose entinostat PO on days 1, 8, and 15, and pembrolizumab intravenously (IV) over 30 minutes on day 1 of cycle 2 and cycles thereafter. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve an objective response or maintain a stable disease (SD) status after the first 4 cycles may continue to receive entinostat and pembrolizumab for up to 1 year.

After completion of study treatment, patients are followed up monthly for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed myelodysplastic syndrome (MDS) diagnosis (regardless of initial International Prognostic Scoring System [IPSS] risk category) or oligoblastic acute myeloid leukemia (AML) with 21-30% bone marrow (BM) blasts in whom DNMTi have failed; patients who have developed AML after DNMTi therapy can be enrolled as long as they have initiated DNMTi therapy while they were in the MDS or oligoblastic AML (20-30% BM blasts) phase and the study chair agrees; failure of DNMTis is defined as: failure to achieve a complete response (CR), partial response (PR) or hematologic improvement (HI) after at least 4 cycles of DNMTi or progressed after such therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Calculated creatinine clearance by Modification of Diet in Renal Disease (MDRD) (CrCl) >= 60 ml/min/1.73 squared meter
* Total bilirubin =< 2.0 mg/dL unless due to Gilbert's syndrome, hemolysis, or ineffective hematopoiesis
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x upper limit of normal (ULN)
* Females of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to start of first cycle of therapy
* Patients must have no clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS leukemia
* Patients must have no serious or uncontrolled medical conditions
* The effects of entinostat and MK-3475 (pembrolizumab) on the developing human fetus are unknown; for this reason, women of child-bearing potential and men who are sexually active with women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men who are sexually active with women of childbearing potential, treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of entinostat and MK3475 (pembrolizumab) administration
* Ability to understand and the willingness to sign a written informed consent document
* Patients, who relapsed 6 months after bone marrow transplant and have no evidence of active graft versus host disease and are off systemic immunosuppressant medications for at least 2 months and have received hypomethylating agents (HMA) therapy before or after transplant and meet other eligibility criteria of progression after at least 4 months of DNMTi therapy, are eligible to be enrolled in this clinical trial
* Patients who are human immunodeficiency virus (HIV) positive may participate IF they meet the following eligibility requirements:

  * Must be on an effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
  * They must have a CD4 count of greater than 250 cells/mcL
  * They must not be receiving prophylactic therapy for an opportunistic infection

Exclusion Criteria:

* Any patients eligible for allogeneic stem cell transplantation (allo-SCT) and willing to undergo allo-SCT as determined at time of screening for trial; patients who are ineligible or not interested in undergoing allo-SCT will be eligible for the trial
* Any serious medical condition, uncontrolled intercurrent illness (e.g., active infection, symptomatic congestive heart failure [CHF], unstable angina, cardiac arrhythmias, laboratory abnormalities, or psychiatric illness and/or biopsychosocial conditions that may limit compliance
* Patients with known active cancers who are on therapy for those cancers at time of screening
* Patients with a known positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection might be enrolled if the viral load by polymerase chain reaction (PCR) is undetectable with/without active treatment
* Pregnant or breast feeding females (lactating females must agree not to breast feed while taking the study drugs)
* Use of any other experimental drug or therapy within 21 days of baseline - patients who have had chemotherapy or radiotherapy within 4 weeks of entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Known hypersensitivity to MK-3475 (pembrolizumab) or history of allergic reactions to compounds of similar chemical or biologic composition to anti-PD1 or PD-L1 antibodies or entinostat
* Prior treatment with any anti-PD-1 blocking therapies or histone deacetylase inhibitors (HDACi), or anti-CTLA-4 antibody, CD137 agonist or other immune activating therapy such as anti-CD 40 antibody within the last 3 months of enrollment in the study
* Any history of active or severe autoimmune disease: inflammatory bowel disease, including ulcerative colitis and Crohn's disease, rheumatoid arthritis, systemic progressive scleroderma, systemic lupus erythematosus, autoimmune vasculitis (e.g., Wegener's granulomatosis), CNS or motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre syndrome, myasthenia gravis, multiple sclerosis); patients with hypothyroidism with stable hormone replacement therapy dosing are allowed on study
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2025-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amer M Zeidan, Principal Investigator — Yale University Cancer Center LAO
Locations (19):
- United States (19):
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Bewersdorf JP, Shallis RM, Sharon E, Park S, Ramaswamy R, Roe CE, Irish JM, Caldwell A, Wei W, Yacoub A, Madanat YF, Zeidner JF, Altman JK, Odenike O, Yerrabothala S, Kovacsovics T, Podoltsev NA, Halene S, Little RF, Piekarz R, Gore SD, Kim TK, Zeidan AM. A multicenter phase Ib trial of the histone deacetylase inhibitor entinostat in combination with pembrolizumab in patients with myelodysplastic syndromes/neoplasms or acute myeloid leukemia refractory to hypomethylating agents. Ann Hematol. 2024 Jan;103(1):105-116. doi: 10.1007/s00277-023-05552-4. Epub 2023 Dec 1. PMID 38036712

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Entinostat, Pembrolizumab) Dose Level 1; Treatment (Entinostat, Pembrolizumab) Dose Level 2: Patients receive lower dose entinostat PO on days 1 and 8 or higher dose entinostat PO on days 1, 8, and 15, and pembrolizumab IV over 30 minutes on day 1 of cycle 2 and cycles thereafter. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve an objective response or maintain a SD status after the first 4 cycles may continue to receive entinostat and pembrolizumab for up to 1 year.
  Entinostat: Given PO
  Pembrolizumab: Given IV
Period: Overall Study
Arm/Group | Treatment (Entinostat, Pembrolizumab) Dose Level 1 | Treatment (Entinostat, Pembrolizumab) Dose Level 2
Started | 22 | 6
Completed | 16 | 3
Not Completed | 6 | 3
Not completed — Death | 2 | 1
Not completed — Physician Decision | 4 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Entinostat, Pembrolizumab) Dose Level 2: Patients receive lower dose entinostat PO on days 1 and 8 or higher dose entinostat PO on days 1, 8, and 15, and pembrolizumab IV over 30 minutes on day 1 of cycle 2 and cycles thereafter. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve an objective response or maintain a SD status after the first 4 cycles may continue to receive entinostat and pembrolizumab for up to 1 year.
  Entinostat: Given PO
- Total: Total of all reporting groups
Arm/Group | Treatment (Entinostat, Pembrolizumab) Dose Level 1 | Treatment (Entinostat, Pembrolizumab) Dose Level 2 | Total
Number analyzed (Participants) | 22 | 6 | 28
Age, Continuous [Median (Full Range); unit: years] | 74 [57 to 86] | 71 [59 to 80] | 73.5 [57 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 17 | 3 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 20 | 6 | 26
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 20 | 5 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 22 | 6 | 28
ECOG performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) scale range: 0-5. 0: Fully active;1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; 4: Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; 5: Dead.
  Participants
    0 | 4 | 0 | 4
    1 | 16 | 3 | 19
    2 | 2 | 3 | 5
Disease [Count of Participants; unit: Participants]
  acute myeloid leukemia (AML) | 3 | 0 | 3
  myelodysplastic syndromes/neoplasms (MDS) | 19 | 6 | 25
Number prior lines of therapy [Median (Full Range); unit: prior therapy lines] | 1 [1 to 4] | 1.5 [1 to 4] | 1 [1 to 4]
Prior Therapy Types [Count of Participants; unit: Participants] — Frequency of participant prior therapy types.
  Participants
    Prior HMA | 22 | 6 | 28
    Azacitidine | 16 | 6 | 22
    Decitabine | 8 | 1 | 9
    HMA combination | 4 | 0 | 4
    ASTX727 | 1 | 0 | 1
    Prior allo-HCT (%) | 0 | 1 | 1
    ≥3 lines of therapy | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Entinostat Given in Combination With Pembrolizumab
Description: Toxicities will be tabulated and graded according to the Common Terminology Criteria for Adverse Events version 5. Dose-limiting toxicities will be assessed after the first 2 cycles of combined therapy. Presented are the counts of participants that experienced DLT in the period up to 42 days.
Time Frame: Up to 42 days
Population: 13 participants were eligible for dose escalation.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Entinostat, Pembrolizumab) Dose Level 1 | Treatment (Entinostat, Pembrolizumab) Dose Level 2
Number analyzed (Participants) | 7 | 6
Participants | 1 | 2

2. Secondary Outcome: Overall Response Rate (Complete Response [CR], Partial Response [PR], Hematologic Improvement [HI])
Description: Will be defined by the modified International Working Group 2006. Rates of CR, PR and HI will be summarized separately by cohort and reported with an exact 95% confidence interval. Upon results entry- best response to combination therapy (number of patients [%]; response assessment after 3 cycles) is presented as counts of the best response.
Time Frame: Up to 6 months after the last dose of entinostat in combination with pembrolizumab ((treatment period: Up to 3, 21-day cycles)
Population: All those enrolled.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Entinostat, Pembrolizumab) DL1; Treatment (Entinostat, Pembrolizumab) DL2: Patients receive lower dose entinostat PO on days 1 and 8 or higher dose entinostat PO on days 1, 8, and 15, and pembrolizumab IV over 30 minutes on day 1 of cycle 2 and cycles thereafter. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve an objective response or maintain a SD status after the first 4 cycles may continue to receive entinostat and pembrolizumab for up to 1 year.
  Entinostat: Given PO
  Pembrolizumab: Given IV
Arm/Group | Treatment (Entinostat, Pembrolizumab) DL1 | Treatment (Entinostat, Pembrolizumab) DL2
Number analyzed (Participants) | 22 | 6
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 0 | 0
  Stable Disease (SD) | 8 | 3
  Progressive Disease (PD) | 5 | 0
  marrow Complete response (mCR) | 2 | 0
  Not evaluable | 6 | 3
  Hematologic Improvement (HI) Neutrophils | 1 | 0

3. Secondary Outcome: Median Progression-free Survival
Description: Median progression-free survival (PFS) is being reported as the median time with the full range. The outcome was updated at the time of results entry to include the correct presentation of the data and the updated time frame for longest PFS follow up time.
Time Frame: Assessed for up to 10 months after the last dose of entinostat in combination with pembrolizumab (treatment period: Up to 3, 21-day cycles)
Population: All participants
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Entinostat, Pembrolizumab) Dose Level 1 | Treatment (Entinostat, Pembrolizumab) Dose Level 2
Number analyzed (Participants) | 22 | 6
months | 3.45 [0.5 to 9.4] | 3.68 [0.9 to 8.8]

4. Other Pre Specified Outcome: Median Response Duration for Responders
Description: Median response duration for responders will be determined.
Time Frame: Up to 6 months after the last dose of entinostat in combination with pembrolizumab
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Median Time of Progression to Acute Myeloid Leukemia
Description: Median time of progression to acute myeloid leukemia will be determined.
Time Frame: Up to 6 months after the last dose of entinostat in combination with pembrolizumab
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Median Overall Survival
Description: Will be reported with a 95% confidence interval.
Time Frame: From start of study to death, assessed for up to 6 months after the last dose of entinostat in combination with pembrolizumab
Reporting Status: Not Posted

7. Other Pre Specified Outcome: 1-year Overall Survival
Description: Will be reported with a 95% confidence interval.
Time Frame: From start of study to death, assessed for up to 1 year
Reporting Status: Not Posted

8. Other Pre Specified Outcome: 2-year Overall Survival
Description: Will be reported with a 95% confidence interval.
Time Frame: From start of study to death, assessed for up to 2 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Dynamic Quantitative Change in Proportion of Myeloid-derived Suppressor Cells (MDSCs) in Bone Marrow With Combined Therapy, Assessed by Flow Cytometry
Description: Will correlate with any observed clinical responses. Will be estimated using mixed effects models to take into account the within-patient correlation. Likelihood ratio tests will be performed to confirm if random intercepts and slopes are necessary in the model. The fixed effect for change in MDSCs over time will be evaluated for significance. The variability in the rate of change in MDSCs across patients will also be examined. The association between the clinical outcome and a meaningful reduction in MDSCs, which will be defined after a review of the data, will be assessed with the chi-square test. The quantity of MDSCs at baseline and during treatment as continuous variables can also be compared between responding and non-responding patients using a t-test or Mann-Whitney U-Test, if more appropriate.
Time Frame: Baseline up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 4 months following treatment (treatment period: Up to 3, 21-day cycles), All-Cause Mortality was assessed up to 10 months after the last dose.
Arm/Group | Treatment (Entinostat, Pembrolizumab) Dose Level 1 | Treatment (Entinostat, Pembrolizumab) Dose Level 2
All-Cause Mortality (participants affected / at risk) | 4/22 | 2/6
Serious Adverse Events (participants affected / at risk) | 12/22 | 5/6
Other Adverse Events (participants affected / at risk) | 22/22 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Entinostat, Pembrolizumab) Dose Level 1 (N=22) | Treatment (Entinostat, Pembrolizumab) Dose Level 2 (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 1 (1) | 0 (0)
Mixed shock (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Immunotherapy -induced pneumonitis (Immune system disorders) | 1 (1) | 0 (0)
Blood infection (Infections and infestations) | 1 (1) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 4 (4) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Disease Progression (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Entinostat, Pembrolizumab) Dose Level 1 (N=22) | Treatment (Entinostat, Pembrolizumab) Dose Level 2 (N=6)
Anemia (Blood and lymphatic system disorders) | 11 (38) | 3 (8)
blood in sputum (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hematemesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
white blood cell increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
hypovolemia (Cardiac disorders) | 0 (0) | 1 (1)
mitral regurgitation (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve regurgitation (Cardiac disorders) | 0 (0) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
volume overload (Cardiac disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid Nodule (Endocrine disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Subconjunctival Hemmorhage (Eye disorders) | 1 (1) | 0 (0)
Subjuntival Hemmorhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barrett's esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 8 (10) | 6 (10)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (5) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 8 (10) | 5 (7)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3)
altered mental status (General disorders) | 1 (1) | 0 (0)
Chest pressure (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 2 (2)
deconditioning (General disorders) | 1 (1) | 0 (0)
decreased appetite (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 4 (4) | 4 (4)
Fatigue (General disorders) | 12 (21) | 6 (9)
Fever (General disorders) | 4 (4) | 4 (5)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
heat in palms (General disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (2) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (3)
pain at biopsy site (General disorders) | 0 (0) | 1 (1)
Post biopsy pain (General disorders) | 1 (1) | 0 (0)
runny nose (General disorders) | 1 (1) | 0 (0)
Soreness (lower back) (General disorders) | 0 (0) | 1 (1)
soreness lower back (General disorders) | 0 (0) | 1 (1)
swelling at port placement site (General disorders) | 0 (0) | 1 (1)
Tooth Loss (General disorders) | 1 (1) | 0 (0)
failure to thrive (Immune system disorders) | 1 (1) | 0 (0)
Recurrent ovarian cancer (Immune system disorders) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Oral Thrush (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
decreased mobility (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scrotal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 3 (5)
Alkaline phosphatase increased (Investigations) | 2 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (5) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 3 (3) | 2 (2)
hyperphosphatemia (Investigations) | 0 (0) | 1 (1)
hyponatremia (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 1 (5) | 0 (0)
Lymphocyte count decreased (Investigations) | 7 (27) | 1 (2)
Lymphocyte count increased (Investigations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 12 (55) | 3 (8)
Platelet count decreased (Investigations) | 15 (74) | 4 (13)
Weight loss (Investigations) | 2 (2) | 2 (6)
white blood cell count increased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 8 (26) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 7 (7) | 2 (4)
cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (6)
Diaphoresis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (8) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (8) | 3 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (17) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 5 (8) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 7 (18) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Generalized body aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4)
muscle cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
muscle pain (right leg) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (4)
right shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 3 (5)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
sensory change (warmth in hands and feet) (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (2)
Chronic kidney disease (Renal and urinary disorders) | 2 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anasarca (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 5 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (2)
mid lung infiltrate (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Pulmonary Aspergillosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
suspected pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
throat burning (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abrasion (left knee) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bilateral Leg Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema - hands (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Excoriation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
mouth sores (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pallor (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechial rash, forearms, easy bruisability (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
wound (right femoral) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bi-lateral leg swelling (Vascular disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT02936752/Prot_SAP_000.pdf